CLINICAL TRIAL: NCT05042440
Title: A Phase 1, Single-Site, Open-Label Study to Assess Pharmacokinetics of Efanesoctocog Alfa (BIVV001), Standard Half-Life and Extended Half-Life FVIII After Each Single Intravenous Injection in a Fixed Sequence, in Previously Treated Adults With Severe Hemophilia A
Brief Title: Pharmacokinetic Assessment of Standard Half-Life (SHL) FVIII, Extended Half-Life (EHL) FVIII, and Efanesoctocog Alfa (BIVV001) in Severe Hemophilia A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PKM17085; 2021-000228-37 (EudraCT Number); U1111-1256-9661 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-08-12; First posted 2021-09-13 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — BIVV001; F8 protein, human; Factor VIII; BAX 855

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- efanesoctocog alfa (BIVV001) (Experimental): Each participant will be sequentially dosed with three single intravenous (IV) doses of first rFVIII (Advate®), second Polyethylene Glycol (PEG)-rFVIII (Adynovi® or Adynovate®), and lastly, BIVV001
  Interventions: Drug: Efanesoctocog alfa; Drug: Octocog alfa; Drug: Rurioctocog alfa pegol

INTERVENTIONS:
Drug: Efanesoctocog alfa — Solution for injection Intravenous
  Other Names: BIVV001
Drug: Octocog alfa — Solution for injection Intravenous
  Other Names: Advate®
Drug: Rurioctocog alfa pegol — Solution for injection Intravenous
  Other Names: Adynovi®

SUMMARY:
Primary objective

• To assess the half-life of BIVV001, Standard Half-Life (SHL) rFVIII and Extended Half-Life (EHL) rFVIII after a single intravenous (IV) injection

Secondary objectives

* To characterize additional pharmacokinetic (PK) parameters of BIVV001, SHL rFVIII and EHL rFVIII after a single IV injection
* To evaluate the safety and tolerability of a single IV injection of BIVV001

DETAILED DESCRIPTION:
This is a Phase 1, single center, open-label, sequential treatment, 3-period fixed sequence study to assess PK profiles of BIVV001, SHL and EHL rFVIII after a single IV injection in male, previously treated patients, 18-65 years of age, with severe hemophilia A (defined as <1 IU/dL [<1%] endogenous FVIII).

The expected duration of the study is up to approximately 67 days including

* Screening and washout up to 28 days,
* Advate® dosing, PK sampling, including washout: approximately 4 days,
* Adynovi® dosing and PK sampling, including washout: approximately 7 days,
* BIVV001 dosing and PK sampling: approximately 14 days, Remainder of Safety Observation Period: approximately 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A, defined as <1 IU/dL (<1%) endogenous FVIII activity.
* Previous treatment for hemophilia A, defined as at least 150 days documented prior exposure to any recombinant and/or plasma-derived FVIII and/or cryoprecipitate products at Day 1.
* Platelet count ≥100,000 cells/µL at Screening.
* A participant known to be human immunodeficiency virus (HIV) antibody positive, either previously documented or identified from screening assessments, must have the following results prior to enrollment. (CD4 lymphocyte count >200 cells/mm³ - Viral load of <400 copies/mL).

Exclusion Criteria:

* Any concurrent clinically significant liver disease that, in the opinion of the Investigator, would make the participant unsuitable for enrollment. This may include, but is not limited to cirrhosis, portal hypertension, and acute hepatitis.
* Serious active bacterial, fungal or viral infection (other than chronic hepatitis or HIV) present within 30 days of Screening.
* Other known coagulation disorder(s) in addition to hemophilia A.
* History of hypersensitivity or anaphylaxis associated with any FVIII product.
* History of a positive inhibitor test defined as ≥0.6 BU/mL, or any value greater than or equal to the lower sensitivity cut-off for laboratories with cut-offs for inhibitor detection between 0.7 and 1.0 BU/mL, or clinical signs or symptoms of decreased response to FVIII administrations. Family history of inhibitors will not exclude the participant.
* Positive inhibitor result, defined as ≥0.6 BU/mL at Screening.
* Major surgery within 8 weeks of Screening.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Half-life of BIVV001 | BIVV001 period: Predose, and post-dose from 0.17 hr to 336 hr, and at day 28
Half-life of SHL rFVIII | Advate® period: Predose, and post-dose from 0.17 hr to 72 hr
Half-Life of EHL rFVIII | Adynovi® period: Predose, and post-dose from 0.17 hr to 120 hr

SECONDARY OUTCOMES:
Assessment of pharmacokinetic (PK) parameter : maximum activity (Cmax) | Predose of each period, 0.17 hr to 72 hr for Advate® ; 0.17 hr to 120 hr for Adynovi® ; 0.17 hr to 336 hr and at day 28 for BIVV001
Assessment of PK parameter : clearance (CL) | Predose of each period, 0.17 hr to 72 hr for Advate® ; 0.17 hr to 120 hr for Adynovi® ; 0.17 hr to 336 hr and at day 28 for BIVV001
Assessment of PK parameter : volume of distribution at steady state (Vss) | Predose of each period, 0.17 hr to 72 hr for Advate® ; 0.17 hr to 120 hr for Adynovi® ; 0.17 hr to 336 hr and at day 28 for BIVV001
Assessment of PK parameter : area under the activity time curve extrapolated to infinity (AUC∞) | Predose of each period, 0.17 hr to 72 hr for Advate® ; 0.17 hr to 120 hr for Adynovi® ; 0.17 hr to 336 hr and at day 28 for BIVV001
Assessment of PK parameter : mean residence time (MRT) | Predose of each period, 0.17 hr to 72 hr for Advate® ; 0.17 hr to 120 hr for Adynovi® ; 0.17 hr to 336 hr and at day 28 for BIVV001
Assessment of PK parameter : incremental recovery (IR) | Predose of each period, 0.17 hr to 72 hr for Advate® ; 0.17 hr to 120 hr for Adynovi® ; 0.17 hr to 336 hr and at day 28 for BIVV001
Number of participants with Adverse events (AE), serious AEs and treatment-emergent AEs (TEAEs) | From Day 1 up to 28 days after administration of BIVV001 (total 39 days including Advate® and Adynovi® period)
Development of inhibitors (neutralizing antibodies directed against FVIII) | Advate® period: Pre-dose; Adynovi® period: Pre-dose; BIVV001 period: Pre-dose and at day 14 and 28 after administration.
  Number of participants with development of inhibitors

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences and Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number :1000001, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Background] Lissitchkov T, Willemze A, Jan C, Zilberstein M, Katragadda S. Pharmacokinetics of recombinant factor VIII in adults with severe hemophilia A: fixed-sequence single-dose study of octocog alfa, rurioctocog alfa pegol, and efanesoctocog alfa. Res Pract Thromb Haemost. 2023 May 13;7(4):100176. doi: 10.1016/j.rpth.2023.100176. eCollection 2023 May. PMID 37538505
- See also: PKM17085 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25325&tenant=MT_SNY_9011